CLINICAL TRIAL: NCT00222209
Title: Implicit Learning, Comorbidity and Stress Vulnerability in Chronic Functional Pain Syndromes
Brief Title: Clinical Study on Implicit Learning, Comorbidity and Stress Vulnerability in Chronic Functional Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: German Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: DFG HO 904/11-3,4
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2006-08-03 (Estimated); Status verified 2005-09

CONDITIONS: Fibromyalgia; Irritable Bowel Syndrome
Keywords: Experimental study; chronic pain; operant learning; comorbidity; stress; Fibromyalgia w visceral hypersensitivity; Fibromyalgia w/o visceral hypersensitivity
MeSH Terms: conditions — Fibromyalgia; Irritable Bowel Syndrome; Chronic Pain

INTERVENTIONS:
Behavioral: Experimental heat pain model

SUMMARY:
The project investigates on the role of pain avoidance, comorbidity and stress response for the development of chronic somatic and visceral pain. We, the researchers at University Hospital Mannheim, assume that implicit operant learning of pain sensitization is a central mechanism of the process of pain becoming chronic, which is augmented by fear and by avoidance behaviour. Somatic and psychological comorbidity as well as stress factors are further promoting factors in chronic pain development.

DETAILED DESCRIPTION:
Study 1: Implicit operant learning of sensitization and habituation in an experimental heat pain model will be investigated and compared in healthy controls, chronic pain patients with fibromyalgia, with and w/o visceral pain.

Study 2: Functional imaging of implicit operant learning of sensitization and habituation in an experimental heat pain model (same subgroups as in study 1).

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia according to American College of Rheumatology (ACR) criteria
* Visceral hypersensitivity according to ROME criteria
* Chronic pain according to International Association for the Study of Pain (IASP) criteria

Exclusion Criteria:

* Abnormal quantitative sensory testing
* Psychiatric or neurological anamnesis, except fear and depression
* Acute major depression
* Substance abuse

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64
Dates: Start 2005-09; Study Completion 2007-11

CONTACTS AND LOCATIONS:
Overall Officials: Rupert Hoelzl, Prof. Dr. phil., Study Director — University of Mannheim; Hans-Joachim Bender, Prof. Dr. med. rer. nat., Study Director — Universitätsmedizin Mannheim; Lothar-Rudi Schad, Prof. Dr. rer. nat., Study Director — German Cancer Research Centre Heidelberg
Locations (1):
- University of Mannheim - Otto-Selz-Institute, Mannheim, Germany

REFERENCES:
- [Background] Holzl R, Kleinbohl D, Huse E. Implicit operant learning of pain sensitization. Pain. 2005 May;115(1-2):12-20. doi: 10.1016/j.pain.2005.01.026. PMID 15836965
- [Background] Kleinbohl D, Holzl R, Moltner A, Rommel C, Weber C, Osswald PM. Psychophysical measures of sensitization to tonic heat discriminate chronic pain patients. Pain. 1999 May;81(1-2):35-43. doi: 10.1016/s0304-3959(98)00266-8. PMID 10353491